CLINICAL TRIAL: NCT02424136
Title: PEAnut Anaphylaxis Predictors
Acronym: PEAAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Hunter Children's Hospital (Other)
Collaborators: Hunter Medical Research Institute, Australia (Unknown); University of Newcastle, Australia (Other); Thrasher Research Fund (Other); Hunter Childrens Research Foundation, Australia (Unknown); Aerocrine AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEAAP (14/12/12/4.12)
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Peanut Hypersensitivity; Anaphylaxis
MeSH Terms: conditions — Peanut Hypersensitivity; Anaphylaxis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entire group (Other): Children aged 2-17 years with suspected peanut allergy who require peanut food challenge to confirm clinical allergy, will be recruited for the study. They will undergo a preceding questionnaire, peanut skin prick testing, spirometry, fraction of exhaled nitric oxide (FeNO) measurement, serum peanut and Ara h2 specific immunoglobulin E (sIgE) antibodies, and collection of blood biomarker prior to food challenge. The primary endpoint will be anaphylaxis at open label peanut challenge, with the primary exposure of interest will be the serum biomarker.
  Interventions: Other: Questionnaire; Other: Peanut Skin prick test; Other: Fraction of exhaled nitric oxide; Other: Spirometry; Other: Serum Peanut and Ara h2 specific immunoglobulin E; Other: Collection of blood biomarker; Other: Peanut food challenge

INTERVENTIONS:
Other: Questionnaire — 5 minute questionnaire focused on symptoms of allergic disease
Other: Peanut Skin prick test — Skin prick testing with peanut antigen, according to ASCIA Skin Prick testing manual
Other: Fraction of exhaled nitric oxide — Measurement of exhaled nitric oxide, according to American Thoracic Society/ European Thoracic Society (ATS/ERS) standardised procedures (Not required for those age less than 6 years).
Other: Spirometry — Measurement of lung flows/volumes, according to ATS/ERS standardised procedures (Not required for those age less than 6 years).
Other: Serum Peanut and Ara h2 specific immunoglobulin E — Peanut and Ara h2 specific IgE antibodies
Other: Collection of blood biomarker — Correlation of blood biomarker levels in patients with successful or unsuccessful peanut food challenge
Other: Peanut food challenge — Open label peanut challenge conducted according to ASCIA's peanut challenge protocol and PRACTALL consensus report

SUMMARY:
Peanut allergy can be life-threatening. Current diagnostic techniques for peanut allergy have high sensitivity, but not high specificity. This clinical trial will test the validity of a novel blood biomarker (compared with current testing) as a diagnostic predictor of anaphylaxis to peanut.

DETAILED DESCRIPTION:
Children aged 2-17 years with suspected peanut allergy will be invited to participate in the study.

They will have a questionnaire, a skin prick test to peanut, 2 breathing tests (spirometry and fraction of exhaled nitric oxide (FeNO)), and a blood test (specific peanut antibodies, allergic immune responses - including the novel blood biomarker - and genetic testing to identify novel potential molecular and genetic markers of food allergy in the future. The genetic testing component will be optional). The breathing test is not required for those under 6 years.

The final step is an open label peanut food challenge with incremental doses of peanut, (routine practise) as per the Australasian Society of Clinical Immunology and Allergy (ASCIA) food challenge protocol.The endpoints in the food challenge will be signs of allergy or anaphylaxis as per PRACTicing ALLergology (PRACTALL) consensus report for oral food challenges OR completion of the ASCIA food challenge protocol.

Outcome: The primary outcome of the project is to confirm that a novel blood biomarker has a higher diagnostic accuracy as compared to current best testing in predicting anaphylaxis at open label peanut challenge.

Secondary outcome: Will be to determine the value of the biomarker, FeNO and Ara h2 specific Immunoglobulin E (sIgE) (individually and in combination) at predicting anaphylaxis or clinical allergy at open label peanut challenge.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 - 17 years with an allergy to peanut and require peanut challenge to confirm peanut allergy.

Exclusion Criteria:

* Children with Peanut Skin Prick Test (SPT) wheal size greater than 10mm as these children are likely to have clinical peanut allergy (no clinical indication for food challenge).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Blood biomarker predicting anaphylaxis at peanut food challenge | At completion of peanut food challenge
  The primary outcome of the project is to confirm that a novel blood biomarker has a higher diagnostic accuracy as compared to current best testing in predicting anaphylaxis at open label peanut challenge.

SECONDARY OUTCOMES:
Blood biomarker in combination with FeNO, and/or Ara h2 sIgE predicting anaphylaxis at peanut food challenge | At completion of peanut food challenge
  The secondary outcome will be to determine the value of the biomarker, FeNO and Ara h2 sIgE (individually and in combination) at predicting anaphylaxis or clinical allergy at open label peanut challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Mattes, MD, Principal Investigator — John Hunter Children's Hospital, Australia
Locations (1):
- John Hunter Children's Hospital, New Lambton, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Derived] Percival E, Bhatia R, Preece K, McEvoy M, Collison A, Mattes J. Change in exhaled nitric oxide during peanut challenge is related to severity of reaction. Allergy Asthma Clin Immunol. 2020 Jul 21;16:64. doi: 10.1186/s13223-020-00464-8. eCollection 2020. PMID 32834829
- See also: ASCIA Skin prick testing for the diagnosis of allergic disease. A manual for practitioners. — https://www.allergy.org.au/images/stories/pospapers/ASCIA_SPT_Manual_March_2016.pdf